CLINICAL TRIAL: NCT04113265
Title: Aesthetic Performance and Tolerance Evaluation of an Injective Intradermal Treatment for the Inner Thighs, Knees and Arms
Brief Title: Aesthetic Performance of an Injective Treatment for the Inner Thighs, Knees and Arms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derming SRL (Other)
Responsible Party: Principal Investigator, Adele Sparavigna, Principal Investigator, Derming SRL
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E0719
Record Dates: First submitted 2019-10-01; First posted 2019-10-02 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Skin Flaccidity Inner Thighs Knees Arms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SUNEKOS ® Body (Experimental): The 1st treatment was performed during T0 visit, after the basal evaluations planned by the study procedure and repeated 3 more times with an interval of 1 week (T2i, T3i and T4i).
  Interventions: Device: SUNEKOS ® Body

INTERVENTIONS:
Device: SUNEKOS ® Body — SUNEKOS ® Body is a medical device (class III). The study product was injected at level of the inner thighs, knees and arms by needle (29 G) using the interstitial fluid technique (IFT)

SUMMARY:
The objective of this study is to investigate the efficacy of the "SUNEKOS® Body" in woman aged 40-65 years with skin flaccidity of the inner thighs, knees and arms.

ELIGIBILITY:
Inclusion Criteria:

* female sex;
* age 40-65 years;
* asking for inner thighs, knees and arms laxity restoration;
* available and able to return to the study site for the post-procedural follow-up examinations;
* accepting to not change their habits regarding food, physical activity, cosmetic and cleansing products for the body;
* accepting not to expose their body to strong UV irradiation (UV session, or sun bathes) during the entire duration of the study, without appropriate sun protection;
* accepting to sign the informed consent form.

Exclusion Criteria:

* Pregnancy;
* lactation;
* smokers;
* alcohol abuse and/or drug use;
* subjects not in menopause who do not use adequate contraceptive precautions in order to avoid pregnancies during the study;
* subjects not in menopause who do not accept to perform the pregnancy test at T0 (before the 1st aesthetic procedure) and at T4i (before the last injection treatment execution);
* Body Mass Index (BMI) variation (± 1) during the study period;
* performing skin treatments for knee, thighs and arms aesthetic correction (carboxytherapy injections, body lifting, laser, infrared light, bipolar radiofrequency, vacuum and mechanical massage) in the 6 months prior to the study start;
* aesthetic surgical procedure on knee, thighs and arms in the past;
* change in the normal habits regarding food, physical activity, cosmetic products and cleansing for the body during the month preceding the test;
* sensitivity to the test product or its ingredients (to be assessed by the investigator during the baseline visit);
* subjects whose insufficient adhesion to the study protocol is foreseeable;
* participation in a similar study currently or during the previous 6 months
* Dermatitis;
* presence of cutaneous disease on the tested area, as lesions, scars, malformations;
* recurrent facial/labial herpes;
* clinical and significant skin condition on the test area (e.g. active eczema, psoriasis, severe rosacea, scleroderma, local infections and severe acne).
* Diabetes;
* endocrine disease;
* hepatic disorder;
* renal disorder;
* cardiac disorder;
* pulmonary disease;
* cancer;
* neurological or psychological disease;
* inflammatory/immunosuppressive disease;
* drug allergy.
* Anticoagulants and antiplatelet drugs, anti-histaminic, topic and systemic corticosteroids, narcotic, antidepressant, immunosuppressive drugs (with the except of contraceptive or hormonal treatment starting more than 1 year ago);
* using of drugs able to influence the test results in the investigator opinion.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline of inner arm skin laxity clinical grade | baseline, 48 hours after the last injection procedure, after 8 weeks, after 16 weeks
  Skin laxity clinical grade, according to a visual score from 1 (no flaccidity) to 5 (very severe flaccidity)
Change from baseline of inner arm skin roughness clinical grade | baseline, 48 hours after the last injection procedure, after 8 weeks, after 16 weeks
  Skin roughness clinical grade, according to a visual score from 1 (no roughness) to 5 (very severe roughness)
Change from baseline of inner thigh skin laxity clinical grade | baseline, 48 hours after the last injection procedure, after 8 weeks, after 16 weeks
  Skin laxity clinical grade, according to a visual score from 1 (no flaccidity) to 5 (very severe flaccidity)
Change from baseline of inner thigh skin roughness clinical grade | baseline, 48 hours after the last injection procedure, after 8 weeks, after 16 weeks
  Skin laxity clinical grade, according to a clinical score from 1 (no roughness) to 5 (very severe roughness)
Change from baseline of inner knee skin laxity clinical grade | baseline, 48 hours after the last injection procedure, after 8 weeks, after 16 weeks
  Skin laxity clinical grade, according to a clinical score from 1 (no flaccidity) to 5 (very severe flaccidity)
Change from baseline of inner knee skin roughness clinical grade | baseline, 48 hours after the last injection procedure, after 8 weeks, after 16 weeks
  Skin laxity clinical grade, according to a visual score from 1 (no roughness) to 5 (very severe roughness)
Change from baseline of superficial skin hydration | baseline, 48 hours after the last injection procedure, after 8 weeks, after 16 weeks
  Skin electrical capacitance value was measured mono-laterally on the right or left inner arm, thigh and knee with Corneometer CM825 (Courage - Khazaka, Köln, Germany). The measure of the skin capacitance properties is an indirect expression of its hydration level.
Change from baseline of deep skin hydration | baseline, 48 hours after the last injection procedure, after 8 weeks, after 16 weeks
  Tissue dielectric constant value of superficial and deep skin layers was measured mono-laterally on the right or left inner arm, thigh and knee with MoistureMeterD (Delfin Technologies, Kuopio - Finland)
Change from baseline of skin density | baseline, 48 hours after the last injection procedure, after 8 weeks, after 16 weeks
  A little skin area of about 7 cm2 (at level of inner arm was pinched, in standardized conditions, using a specific device. Because of this "pinch" the skin profile changes depending on cutaneous density; when the skin is slack the "pinch" forms a lot of wrinkles. A picture of the skin pinched was taken thanks to Primos compact portable device (GFMesstechnik); Primos software is able to measure skin principal profilometric parameters.
Change from baseline of photographic documentation | baseline, 48 hours after the last injection procedure, after 8 weeks, after 16 weeks
  2D pictures of the inner arm, thigh and knee

CONTACTS AND LOCATIONS:
Locations (1):
- DERMING, Milan, MI, Italy